CLINICAL TRIAL: NCT03393520
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-design Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Assessment of the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-AVP-786-305; 2017-001339-38 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type
Keywords: Agitation; Dementia of the Alzheimer's type; Alzheimer's disease; AVP-786; Deudextromethorphan hydrobromide; Quinidine sulfate
MeSH Terms: conditions — Psychomotor Agitation; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will be assigned to treatment with placebo capsules administered twice a day over a 12-week period.
  Interventions: Drug: Placebo
- AVP-786; Dose 1 (Experimental): Participants will receive AVP-786 (Dose 1) capsules administered twice a day over a 12-week period.
  Interventions: Drug: AVP-786
- AVP-786; Dose 2 (Experimental): Participants will receive AVP-786 (Dose 2) capsules administered twice a day over a 12-week period.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: Placebo — oral capsules
  Arms: Placebo
Drug: AVP-786 — oral capsules
  Arms: AVP-786; Dose 1; AVP-786; Dose 2

SUMMARY:
This study will be conducted to evaluate the efficacy, safety, and tolerability of AVP-786 compared to placebo, for the treatment of agitation in participants with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of probable Alzheimer's disease (AD) and must have clinically significant, moderate/severe agitation secondary to AD.

This is a multicenter, randomized, double-blind, placebo-controlled, parallel-design study, consisting of 12 weeks of treatment.

Approximately 550 participants will be enrolled at approximately 90 centers worldwide.

Study medication will be administered orally twice-daily from Day 1 through Day 85. Screening will occur within approximately 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease (AD) according to the 2011 National Institute on Aging-Alzheimer's Association (NIA-AA) working groups criteria
* Participants with clinically significant, moderate/severe agitation at the time of screening and for at least 2 weeks prior to baseline that interferes with their daily routine and for which a prescription medication has been indicated, in the opinion of the investigator
* The diagnosis of agitation must meet the provisional consensus definition of agitation in participants with cognitive disorders developed by the International Psychogeriatric Association (IPA) Agitation Definition Work Group.
* A Clinical Global Impression of Severity of Illness scale for Agitation (CGIS-Agitation) score of ≥ 4 (moderately ill) at screening and baseline
* Participants must have a reliable caregiver who is able and willing to comply with study procedures, including not administering any prohibited medications during the course of the study.
* Caregiver who is able and willing to comply with all required study procedures. In order to qualify as a reliable informant (i.e., caregiver) capable of assessing changes in participant's condition during the study, the individual must spend a minimum of 2 hours per day for 4 days per week with the participant.

Exclusion Criteria:

* Participants with dementia predominantly of the non-Alzheimer's type (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia)
* Participants with symptoms of agitation that are not secondary to AD (e.g., secondary to pain, other psychiatric disorder, or delirium)
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participants with myasthenia gravis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score | Baseline; Week 12

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in the Clinical Global Impression of Severity (CGIS)-Agitation Domain Score | Baseline; Week 12

CONTACTS AND LOCATIONS:
Locations (211):
- United States (93):
  - MD First Research #767, Chandler, Arizona
  - Liv Generations of Agritopia / CCT #573, Gilbert, Arizona
  - Liv Generations of Ahwatukee / CCT #784, Phoenix, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - Medical Advancement Center of Arizona #820, Tempe, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - Advanced Research Center, Inc #835, Anaheim, California
  - ATP Clinical Research, Inc #763, Costa Mesa, California
  - Paradigm Clinical Research Centers, Inc., La Mesa, California
  - Sunwise Clinical Research #831, Lafayette, California
  - Torrance Clinical Research Institute, Inc. #826, Lomita, California
  - Rohun Medical Corporation Site #770, Long Beach, California
  - Alliance for Wellness, Inc dba Alliance for Research #789, Long Beach, California
  - Havana Research Institute, Pasadena, California
  - Neurology of Central Florida Rsch Ctr # 803, Altamonte Springs, Florida
  - Negron Research Services / Humanity Clinical Research #766, Aventura, Florida
  - SFM Clinical Research, LLC #563, Boca Raton, Florida
  - Helix Biomedics LLC, Boynton Beach, Florida
  - Bradenton Research Center #834, Bradenton, Florida
  - Clinical Research of Brandon #838, Brandon, Florida
  - ASCLEPES Research Center #806, Brooksville, Florida
  - Beautiful Minds Clinical Research Center #808, Cutler Bay, Florida
  - Science Connections, LLC #814, Doral, Florida
  - ConSalud Medical Research #773, Hialeah, Florida
  - Direct Helpers Research Center # 801, Hialeah, Florida
  - New Med Research Inc #812, Hollywood, Florida
  - Alphab Global Research #793, Jupiter, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Meridien Research - Lakeland Site Site #558, Lakeland, Florida
  - Zynak Clinical Services, Lauderdale Lakes, Florida
  - Adaptive Clinical Research, Inc. Site# 815, Lauderhill, Florida
  - Innovative Clinical Research, Inc Site #819, Lauderhill, Florida
  - Homestead Associates in Research #797, Miami, Florida
  - Premier Clinical Research Institute, Inc. #817, Miami, Florida
  - Central Miami Medical Institute # 798, Miami, Florida
  - Project4Research #774, Miami, Florida
  - City Medical Group RC, Miami, Florida
  - Finlay Medical Research Corp #552, Miami, Florida
  - First Class Medical Services #807, Miami, Florida
  - Miami Jewish Health Systems, Inc. #786, Miami, Florida
  - New Horizon Research Center Site #795, Miami, Florida
  - Reliant Medical Research, LLC #811, Miami, Florida
  - Clinical Research Associates of South Florida, Miami, Florida
  - P&S Research, LLC #805, Miami, Florida
  - Pharmax Research of South Florida, Miami, Florida
  - Research Institute of West Kendall, Miami, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - Agility Medical Research, Inc Site #816, Miami Lakes, Florida
  - Bayside Clinical Research, New Port Richey, Florida
  - Combined Research Orlando #799, Orlando, Florida
  - Innovation Medical Research Center #802, Palmetto, Florida
  - Quantum Laboratories Site #768, Pompano Beach, Florida
  - Neurostudies Inc. Site# 796, Port Charlotte, Florida
  - VICIS Clinical Research Inc. #777, Tampa, Florida
  - Academic Alliance in Dermatology, Tampa, Florida
  - JSV Clinical Research Study, Inc. #829, Tampa, Florida
  - NeuroStudies. Net, LLC, Decatur, Georgia
  - Hawaii Pacific Neuroscience #833, Honolulu, Hawaii
  - DelRicht Research #776, Covington, Louisiana
  - Alzheimer Disease Center #804, Braintree, Massachusetts
  - Neurobehavioral Medicine Group #828, Bloomfield, Michigan
  - Onyx Clinical Research, LLC, Caro, Michigan
  - Oakland Medical Research #762, Troy, Michigan
  - Precise Research Centers Site #765, Flowood, Mississippi
  - Galen Research Site #550, Chesterfield, Missouri
  - Psychiatric Care and Research Center #827, O'Fallon, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Mid Hudson Medical Research, PLLC #836, New Windsor, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Five Towns Neurology PC/Village Site #764, Woodmere, New York
  - The Neurological Institute #843, Charlotte, North Carolina
  - New Hope Clinical Research, Charlotte, North Carolina
  - Insight Clinical Trials LLC #570, Beachwood, Ohio
  - Valley Medical Research Site#788, Centerville, Ohio
  - Osumc #837, Columbus, Ohio
  - NorthStar Medical Research #778, Middleburg Heights, Ohio
  - Onyx Clinical Research, LLC, Youngstown, Ohio
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - Orenda Research & Consulting LLC #840, Oklahoma City, Oklahoma
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Trinity Universal Research Associates Site #821, Carrollton, Texas
  - Texas Neurology #832, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Bio Pharma Informatic LLC Site #822, Houston, Texas
  - Bio Pharma Informatic Inc Site #769, Houston, Texas
  - Katy Neurology #823, Katy, Texas
  - Northpointe Psychiatry #761, Lewisville, Texas
  - Wellness Clinical Research #824, McKinney, Texas
  - PRX Research Site #825, Mesquite, Texas
  - Wasatch Clinical Research, LLC Site #771, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research # 772, Everett, Washington
  - IPC Research, Waukesha, Wisconsin
- Australia (3):
  - Australian Alzheimer's Research Foundation, Nedlands
  - Neuro Trials Victoria Pty Ltd, Noble Park
  - The Alfred Hospital, Parkville
- Bulgaria (12):
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski, Pleven
  - Medical Center Hipokrat-N EOOD, Plovdiv
  - Center for Mental Health - Ruse, Rousse
  - Mental Health Centre Prof.Nikola Shipkovenski #713, Sofia
  - DCC "Sv. Vrach and Sv. Sv. Kuzma and Damian" OOD #710, Sofia
  - First Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Medical Center Stimul, Sofia
  - Medical Center Sveti Naum #707, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska, Sofia
  - Diagnostic-consultative center Mladost-М Varna OOD #711, Varna
  - Medica Plus Medical Center #705, Veliko Tarnovo
  - Mental Health Center Site #712, Vratsa
- Czechia (14):
  - MUDr. Marta Holanová Site# 733, Brno
  - Fakultni Nemocnice u sv. Anny v Brne #722, Brno
  - Clinline Services s.r.0 Psychiatricka ambulance #732, Hostivice
  - Fakultní Nemocnice Hradec Králové #724, Hradec Kralové
  - NeuropsychiatrieHK #729, Hradec Králové
  - Brain-Soultherapy #728, Kladno
  - Supervize #723, Kutná Hora
  - A-Shine s.r.o., Pilsen
  - Ad71 #727, Prague
  - Clintrial #720, Prague
  - INEP Medical s.r.o. Institut Neuropsychiatricke Pece #730, Prague
  - Neurologicka Ambulance - Forbeli #721, Prague
  - Neuropsychiatrie #726, Prague
  - Vestra Clinics #725, Rychnov nad Kněžnou
- France (8):
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre, Caen
  - Centre Hospitalier de Calais, Calais
  - Centre Hospitalier Universitaire Dijon Bourgogn #536, Dijon
  - Centre Hospitalier Universitaire de Nantes - Hôpital Nord Laennec #537, Nantes
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Saint-Étienne - Hôpital Nord #535, Saint-Etienne
  - Centre Hospitalier Universitaire Toulouse - Casselardit Ancely #533, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Hungary (13):
  - Dr. Kenessey Albert Kórház-Rendelőintézet, Balassagyarmat
  - Semmelweis Egyetem Site #595, Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak #586, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - Valeomed Egeszsegugyi es Szolgaltato Kft, Esztergom
  - Petz Aladár Egyetemi Oktató Kórház Site# 594, Győr
  - Dr. Mathe es Tarsa Beteti Tarsasa Site #593, Kalocsa
  - CRU Hungary Egészségügyi és Szolgáltató Korlátolt Felelősségű Társaság, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - PsychoTech #580, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
- Italy (10):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Centro San Giovanni di Dio - Fatebenefratelli, Brescia
  - Università degli studi G.D'Annunzio Chieti Pescara, Chieti
  - Azienda Ospedaliero - Universitaria Careggi #610, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - Azienda Sanitaria Locale di Biella - Nuovo Ospedale degli Infermi, Ponderano
  - Azienda Ospedaliera Sant'Andrea #606, Roma
  - Fondazione Policlinico Tor Vergata #609, Roma
  - Fondazione Santa Lucia - Istituto di Ricovero e Cura a Carattere Scientifico, Roma
- Poland (19):
  - Śródmieście Przychodnia - Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Sensemed, Chorzów
  - Care Clinic #750, Katowice
  - Wielospecjalistyczna Poradnia Lekarska Synapsis #741, Katowice
  - Krakowska Akademia Neurologii #740, Krakow
  - Pratia MCM Kraków #747, Krakow
  - Medycyna Milorzab #743, Lodz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol #757, Nowa Sól
  - Neurologiczny Niepubliczny Zakład Opieki Zdrowotnej, Plewiska
  - Centrum Medyczne HCP, Poznan
  - Solumed Centrum Medyczne #753, Poznan
  - RCMed Oddział Sochaczew #510, Sochaczew
  - Amonaria Indywidualna Specjalistyczna Praktyka Lekarska Agnieszka Remlinger-Molenda #508, Suchy Las
  - Centrum Medyczne Euromedis, Szczecin
  - Ośrodek Alzheimerowski #756, Ścinawa
  - Przychodnia Specjalistyczna Prosen Site#758, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - ClinHouse Centrum Medyczne #755, Zabrze
- South Africa (6):
  - ACF Neurological Services, Cape Town
  - Cape Trial Centre #621, Cape Town
  - Flexivest Fourteen Research Centre #620, Cape Town
  - Apollo Clinical Research #623, Johannesburg
  - Medical and Dental Centre #625, Rosebank
  - Dr. Chisto Carel Coetzee, Umhlanga
- Spain (19):
  - Accellacare Alcobendas #659, Alcobendas, Aocobendas
  - Fundació ACE, Barcelona
  - Fundació Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario Reina Sofia #647, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari de Santa Maria, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda #658, Majadahonda
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca #656, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena #649, Seville
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Complejo Asistencial de Zamora Hospital Virgen de la Concha #652, Zamora
  - Hospital Viamed Montecanal #643, Zaragoza
- United Kingdom (14):
  - MAC Clinical Research - Barnsley Site #671, Barnsley
  - Research Institute for the Care of Older People, Bath
  - Belfast Health and Social Care Trust, Belfast
  - MAC Clinical Research - Blackpool, Blackpool
  - MAC Clinical Research - Cannock #672, Cannock
  - MAC Clinical Research - Leeds, Leeds
  - Re:Cognition Health - London, London
  - South London and Maudsley NHS Foundation Trust, London
  - MAC Clinical Research - Manchester, Manchester
  - Northamptonshire Healthcare NHS Foundation Trust #682, Northampton
  - MAC Clinical Research - Liverpool, Prescot
  - Southern Health NHS Foundation Trust #679, Southampton
  - Avon and Wiltshire Mental Health Partnership NHS Trust, Swindon
  - North West Boroughs Healthcare NHS Foundation Trust #685, Warrington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com